CLINICAL TRIAL: NCT00896272
Title: Adaptation Among Adolescents and Adults With Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909142; 09-HG-N142
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-01-13

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter Syndrome; 47,XXY; XXY
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study aims to understand the impact of living with Klinefelter syndrome (KS) and the factors that contribute to adaptation in adolescents and adults. Individuals with KS may have variable symptoms, including hypogonadism, gynecomastia, learning disabilities, and delay and underdevelopment of secondary sexual characteristics. Perhaps the most challenging symptom of KS is infertility, which seems to be a universal symptom. It is not fully understood how males with KS conceptualize their condition, cope with their diagnosis, and adapt to living with this condition. In this study, Lazarus and Folkman s Transactional Model of Stress and Coping provides a framework for examining coping and adaptation in males with KS. A cross-sectional research design using a quantitative survey will be utilized to examine the relationships among appraisals (illness perceptions and perceived stigma), time elapsed since learning of diagnosis, coping, and adaptation. Adolescents and adults with KS will be recruited from national KS support networks via website postings, email listservs, and printed newsletter postings. Adolescents will also be recruited from a private practice. Participants will have the option to complete an online or paper version of the survey. The main outcome variable is adaptation to living with a KS diagnosis.

DETAILED DESCRIPTION:
This study aims to understand the impact of living with Klinefelter syndrome (KS) and the factors that contribute to adaptation in adolescents and adults. Individuals with KS may have variable symptoms, including hypogonadism, gynecomastia, learning disabilities, and delay and underdevelopment of secondary sexual characteristics. Perhaps the most challenging symptom of KS is infertility, which seems to be a universal symptom. It is not fully understood how males with KS conceptualize their condition, cope with their diagnosis, and adapt to living with this condition. In this study, Lazarus and Folkman s Transactional Model of Stress and Coping provides a framework for examining coping and adaptation in males with KS. A cross-sectional research design using a quantitative survey will be utilized to examine the relationships among appraisals (illness perceptions and perceived stigma), time elapsed since learning of diagnosis, coping, and adaptation. Adolescents and adults with KS will be recruited from national KS support networks via website postings, email listservs, and printed newsletter postings. Adolescents will also be recruited from a private practice. Participants will have the option to complete an online or paper version of the survey. The main outcome variable is adaptation to living with a KS diagnosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Must have Klinefelter syndrome (47,XXY) by self-report.
  2. Must be 14 years or older.

Ages: 14 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2009-05-05; Study Completion 2015-01-13

PRIMARY OUTCOMES:
Adaptation to Klinefelter. The primary research question is to answer how adolescents and adults adapt to Klinefelter syndrome.

SECONDARY OUTCOMES:
Open ended questions will also assess most difficult and best aspects of living with the condition. Follow-up research will be aimed at opportunities for enhancing adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abramsky L, Chapple J. 47,XXY (Klinefelter syndrome) and 47,XYY: estimated rates of and indication for postnatal diagnosis with implications for prenatal counselling. Prenat Diagn. 1997 Apr;17(4):363-8. doi: 10.1002/(sici)1097-0223(199704)17:43.0.co;2-o. PMID 9160389
- [Background] Biesecker BB, Erby L. Adaptation to living with a genetic condition or risk: a mini-review. Clin Genet. 2008 Nov;74(5):401-7. doi: 10.1111/j.1399-0004.2008.01088.x. Epub 2008 Sep 24. PMID 18823383
- [Background] Bender BG, Harmon RJ, Linden MG, Robinson A. Psychosocial adaptation of 39 adolescents with sex chromosome abnormalities. Pediatrics. 1995 Aug;96(2 Pt 1):302-8. PMID 7630689